CLINICAL TRIAL: NCT00188942
Title: Neural Correlates of Emotional Processing in Depressed and Remitted Bipolar and Unipolar Depressed Subjects: An fMRI Investigation
Brief Title: A Neuroimaging Investigation of Brain Activity in Major Depressive Disorder and Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Sidney Kennedy, Principal Investigator, University Health Network, Toronto
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 04-0204-B; CTA Control #095694
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Major Depressive Disorder
Keywords: Magnetic Resonance Imaging; Diagnostic Imaging; Mood Disorders; Major Depressive Disorder; Antipsychotic; Olanzapine; Fluoxetine
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders | interventions — olanzapine-fluoxetine combination; Olanzapine

ARMS (1):
- Fluoxetine + Olanzapine (Active Comparator)
  Interventions: Drug: Fluoxetine+Olanzapine; Drug: Olanzapine; Procedure: Functional Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Fluoxetine+Olanzapine
Drug: Olanzapine
Procedure: Functional Magnetic Resonance Imaging

SUMMARY:
This study employs functional magnetic resonance imaging to compare brain activation patterns during a depressive episode in patients diagnosed with bipolar disorder, major depressive disorder, and a group of healthy control subjects. Depressed patients will be treated with a combination of fluoxetine and olanzapine and undergo MRI scans before, during, and after pharmacotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to further characterize the neural correlates of affective processing in BD and MDD subjects using fMRI. Subjects who meet criteria for a major depressive episode in the context of BD (n=15); MDD (n=15) and a group of psychiatrically unaffected control subjects (CS, n=15) will undergo four fMRI scans while experiencing a temporary mood induction through the presentation of affective imagery from the International Affective Picture System (IAPS). Both BD and MDD subjects will receive the same combination pharmacotherapy to treat the depression, with fMRI data acquired before, and 1, 3, 6 weeks following pharmacotherapy initiation. Positive, negative, and neutral affective visual stimuli will be presented in a blocked design.

Comparison(s): The effects of time and group will be analyzed in factorial models. Regions of interest that demonstrate significant group-by-time interactions will be further correlated with self-report and clinician-rated psychometric indices.

ELIGIBILITY:
Inclusion Criteria: (All three groups)

* age 18-55 years
* satisfactory physical health
* education level and a degree of understanding to communicate effectively with the investigator c
* capable of providing informed consent
* female subjects of childbearing potential, a medically accepted means of contraception.

Additional inclusion criteria for the patient groups include

* DSM-IV-TR criteria for a diagnosis of BD or MDD
* currently meeting criteria for an MDE and
* a Hamilton Depression Rating Scale 17 Item (HDRS-17) score of > 17
* blood indices within normal clinical ranges.

Exclusion Criteria: (All three groups)

* DSM-IV-TR criteria for substance abuse or dependence (except nicotine or caffeine) within the past 6 months
* comorbid neurological or other major psychiatric disorders as defined in the DSM-IV-TR;
* history of neurological trauma resulting in loss of consciousness;
* uncorrected hypothyroidism or hyperthyroidism, including elevated thyroid stimulating hormone (TSH);
* other unstable medical condition;
* female subjects who are pregnant or nursing;

Additional exclusion criteria for the BD and MDD group include:

* prior failure to respond to fluoxetine and olanzapine in combination at adequate dose and duration;
* evidence of serious risk of suicide based on clinician assessment and/or HRSD suicide item > 3;
* course of ECT (electroconvulsive therapy) in the preceding 6 months;
* Young Mania Rating Scale (YMRS) > 7;
* administration of fluoxetine within previous 4 weeks;
* treatment resistance as defined by the failure of two antidepressant trials from dissimilar classes
* Hyperglycemia or diabetes mellitus as defined by a fasting blood glucose value of > 125 mg/dl.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2005-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
MRI Data - Acquired before and 1- 3- and 6- weeks after beginning pharmacotherapy. | 6 weeks
17 Item - Hamilton Depression Rating Scale - Weekly | 6 weeks
Clinical Global Impression - Improvement/Severity - Weekly | 6 weeks
Young Mania Rating Scale - Weekly | 6 weeks

SECONDARY OUTCOMES:
Positive Affect Negative Affect Scale | 6 weeks
Beck Depression Inventory | 6 weeks
State Trait Anxiety Index | 6 weeks
Behavioural Activation/Inhibition Scale | 6 weeks
SexFX Scale | 6 weeks
AMDP-5 Symptom Questionnaire | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H. Kennedy, MD, FRCPC, Principal Investigator — University Health Network, Department of Psychiatry, University of Toronto
Locations (2):
- Canada (2):
  - University Health Network - Toronto General Division, Toronto, Ontario
  - University Health Network - Toronto Western Division, Toronto, Ontario

REFERENCES:
- [Background] Kumari V, Mitterschiffthaler MT, Teasdale JD, Malhi GS, Brown RG, Giampietro V, Brammer MJ, Poon L, Simmons A, Williams SC, Checkley SA, Sharma T. Neural abnormalities during cognitive generation of affect in treatment-resistant depression. Biol Psychiatry. 2003 Oct 15;54(8):777-91. doi: 10.1016/s0006-3223(02)01785-7. PMID 14550677
- [Background] Malhi GS, Lagopoulos J, Ward PB, Kumari V, Mitchell PB, Parker GB, Ivanovski B, Sachdev P. Cognitive generation of affect in bipolar depression: an fMRI study. Eur J Neurosci. 2004 Feb;19(3):741-54. doi: 10.1111/j.0953-816x.2003.03159.x. PMID 14984424
- [Background] Davidson RJ, Irwin W, Anderle MJ, Kalin NH. The neural substrates of affective processing in depressed patients treated with venlafaxine. Am J Psychiatry. 2003 Jan;160(1):64-75. doi: 10.1176/appi.ajp.160.1.64. PMID 12505803